CLINICAL TRIAL: NCT02057107
Title: Randomized Phase II Trial of Stereotactic Body Radiation Therapy (SBRT) With Cetuximab +/- Docetaxel Followed by Adjuvant Cetuximab +/- Docetaxel in Recurrent, Previously-Irradiated Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: SBRT With Cetuximab +/- Docetaxel Followed by Adjuvant Cetuximab +/- Docetaxel in Recurrent, Previously-Irradiated SCCHN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heath Skinner (Other)
Responsible Party: Sponsor-Investigator, Heath Skinner, Medical Director, Dept. of Radiation Oncology and Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 11-112
Record Dates: First submitted 2014-01-30; First posted 2014-02-06 (Estimated); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Previously-Irradiated; Squamous Cell Carcinoma of the Head and Neck Cancer
Keywords: Stereotactic Body Radiation Therapy (SBRT)
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiosurgery; Cetuximab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- SBRT + Cetuximab + Docetaxel followed by Cetuximab + Docetaxel (Other): Previously Treated With Cetuximab - Group A; No Previous Cetuximab - Group C
  Interventions: Radiation: SBRT; Drug: Cetuximab; Drug: Docetaxel
- SBRT + Cetuximab followed by Cetuximab (Other): Previously Treated with Cetuximab - Group B; No Previous Cetuximab - Group D
  Interventions: Radiation: SBRT; Drug: Cetuximab

INTERVENTIONS:
Radiation: SBRT — 8.8-10 Gy per fraction (total: 44-50 Gy)
  Other Names: Radiosurgery; Stereotactic radiosurgery; CyberKnife; True Beam; Trilogy
Drug: Cetuximab — Day -7 (One week prior to commencement of stereotactic radiosurgery):
  Cetuximab, 400 mg/m2
  Days 0 and 8 (The 1st and 2nd week of radiosurgery):
  Cetuximab, 250 mg/m2 Cetuximab, 250 mg/m2 will be given weekly ( following radiosurgery)
  Other Names: Erbitux
Drug: Docetaxel — Days 0 and 8 (The 1st and 2nd week of radiosurgery) Docetaxel, 25 mg/m2 Docetaxel, 25 mg/m2 will be given weekly (following radiosurgery)
  Other Names: Taxotere
  Arms: SBRT + Cetuximab + Docetaxel followed by Cetuximab + Docetaxel

SUMMARY:
The aim of this trial is to examine the addition of docetaxel on disease progression, metastasis and survival of patients otherwise treated with SBRT and cetuximab alone. To better resolve the impact of the experimental treatment the presence/absence of prior cetuximab treatment will be determine before assigning treatment to either cetuximab and SBRT only or cetuximab, SBRT, and docetaxel.

DETAILED DESCRIPTION:
The aim of this trial is to examine the addition of docetaxel on the overall survival of patients otherwise treated with SBRT and cetuximab alone. In addition, we will determine the difference in progression free survival (PFS), the rate of local recurrence (LR) and of distant metastases (DM) across the SBRT and cetuximab + docetaxel arm and the arm receiving SBRT and cetuximab alone. To better resolve the impact of the experimental treatment on PFS, LR, and DM, patients will be stratified by the presence/absence of prior cetuximab treatment and then randomized to either the control arm (cetuximab and SBRT only) or the experimental arm (cetuximab, SBRT, and docetaxel).

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven recurrent squamous cell carcinoma of the head and neck (SCCHN), who has received prior radiotherapy with or without chemotherapy. New primary is allowed if location is in a previously irradiated field. Biopsy is recommended for each recurrence but is not mandated per study. This will be at the discretion of the principal investigator.
* Prior radiation dose of at least 50 Gy.
* Disease confined to locoregional site and can be encompassed in a stereotactic body radiosurgery "portal"
* Tumor must be deemed to be inoperable or unresectable either by clinical or radiographic criteria. These criteria include encasement of great vessels, vertebral invasion or undue peri-operative risk.
* Prior surgery for recurrent or new SCCHN is allowed in previously irradiated patients. A minimum of 4 weeks should elapse between any surgery and treatment on study. However, high-risk pathologic features should be present, such as positive margins, positive lymphadenopathy, perineural or angiolymphatic invasion.
* Karnofsky performance status > 60 (ECOG 0-1)
* Prior treatment with an EGFR Inhibitor is allowed if it was a part of prior curative therapy and was completed at least 30 days prior to commencement of study therapy
* Any number of prior chemotherapy regimens are allowed
* Measurable disease on imaging studies (MRI, CT, PET-CT or physical exam)
* Age > 18
* Estimated life expectancy > 12 weeks
* No prior radiation therapy or chemotherapy within 1 month of study enrollment
* ANC > 1000, PLT>75,000, Serum creatinine<2.5 mg/dL, Bilirubin <1.5 x upper limits of normal (ULN)
* Diabetes must be controlled prior to PET-CT scanning (blood glucose <200 mg/dL)
* Ability to provide written informed consent

Exclusion Criteria:

* Evidence of distant metastasis on upright chest x-ray (CXR), computed tomography (CT) or other staging studies
* Patients in their reproductive age group should use an effective method of birth control. Patients who are breast-feeding, or have a positive pregnancy test will be excluded from the study
* Any co-morbidity or condition of sufficient severity to limit full compliance with the protocol per assessment by the investigator
* Concurrent serious infection
* History of known hypersensitivity to cetuximab, docetaxel or similar agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-07-03 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
1-Year Locoregional Progression-free survival (PFS) | Up to 12 months
  The proportion of previously-irradiated patients treated with SBRT, cetuximab, and/or docetaxel, evaluated by PET/CT per RECIST Criteria v1.1 that do not experience locoregional disease progression within one year. Per RECIST, Progressive Disease is defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s).
Incidence of distant disease | Up to 12 months
  The proportion of patients with distant disease evaluated by PET/CT or CT per RECIST Criteria v1.1. Malignant disease that has spread to other organs or to lymph nodes other than those near the primary tumor. Per RECIST, Progressive Disease is defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s).
Acute toxicities | Up to 3 months after SBRT treatment
  Adverse Events and Serious Adverse Events determined by patient follow up per CTCAE v4.0 criteria.
Late toxicities | From 3 months after SBRT treatment, up to 3 years
  Adverse Events and Serious Adverse Events determined by patient follow up per CTCAE v4.0 criteria.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 12 months
  Incidence of either a confirmed Complete Response (CR) or Partial Response (PR), per RECIST Criteria v1.1. Per RECIST, CR is defined as the disappearance of all target lesions. To be assigned a status of complete response, changes in tumor measurements must be confirmed by repeat assessments performed no less than four weeks after the criteria for response are first met. PR is defined as at least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum longest diameter. To be assigned a status of partial response, changes in tumor measurements must be confirmed by repeat assessments performed no less than four weeks after the criteria for response are first met.
Overall Survival (OS) | Up to 5 years
  Time from the date of randomization to the date of death due to any cause.
University of Washington QOL Assessment Tool (UW-QOL) | Up to 5 years
  The UW-QOL is a patient-reported outcome measure consisting of domains based upon discrete ordinal responses regarding their past 7 days. Scoring is scaled to so that a score of 0 represents the worst possible response, and a score of 100 represents the best possible response. 12 single question domains, these having between 3 and 6 response options that are scaled evenly from 0 (worst) to 100 (best) according to the hierarchy of response. The domains are pain, appearance, activity, recreation, swallowing, chewing, speech, shoulder, taste, saliva, mood and anxiety. Another question asks patients to choose up to three of these domains that have been the most important to them. There are also three global questions, one about how patients feel relative to before they developed their cancer, one about their health-related QOL and one about their overall QOL.
Progression-free Survival (PFS) | Up to 5 years
  Time from the date of entry on study to the date of progression per RECIST Criteria v1.1 or the date of death from any cause. Subjects who are alive and have not progressed will be censored at their last follow-up date. Per RECIST, Progressive Disease is defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s).

CONTACTS AND LOCATIONS:
Overall Officials: David A Clump, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center - Radiation Oncology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No